CLINICAL TRIAL: NCT06058026
Title: Clinical Evaluation of Composite Resins in Class II Cavities
Brief Title: Clinical Comparison of Composite Materials
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Assistan Professor, Recep Tayyip Erdogan University
Other Study IDs: RTEUDHFMKARADAS001
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-02

CONDITIONS: Caries; Dentin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: World Dental Federation criteria (FDI) — Restorations were evaluated with FDI criteria.

SUMMARY:
Universal adhesive solutions have just entered the market, allowing dentists to choose an adhesive strategy based on the needs of patients and clinical situations. Theses adhesives contain a primer/adhesive resin mix in a single bottle for multi-mode etch-and-rinse or self-etch applications. The aim of this study was to evaluate the clinical performance of composite resins with diffent adesive agents on Class II cavities.

DETAILED DESCRIPTION:
This study was a double-blind (evaluator and patient) randomized controlled clinical study with six study groups with an equal allocation. Two composite materials with two universal and one two-step self-etch adhesives were compared in Class II restorations.

The treated patients were called back for controls after one week, six months, and eighteen months. Restorations were evaluated clinically according to modified FDI criteria. In terms of esthetic property, marginal discoloration; in terms of function properties, fracture and retention, and marginal adaptation; in terms of the biological characteristics, post-operative sensitivity, and secondary caries criteria were examined.

Clinical evaluation was performed by two qualified clinicians. Bite-wing radiographs were taken from the patients who were called for controls at 6-moth and 18-month to evaluate the formation of secondary caries.

Differences between adhesives at each time period were evaluated using Fisher's Exact test. The effect of time on restorations was evaluated using the Friedman test (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Individuals without systemic disease
* Individuals with good oral hygiene
* Must be a minimum of one carious defect
* Must be at least 18 years old
* Must have vital teeth in antagonist and proximal contact.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Receiving orthodontic treatment
* Bruxism habit
* Direct or indirect pulp coverage
* Allergy to resin-based products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Teeth with primary caries, including at least one-third of the dentin (MO or DO), were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of class II restorative materials restored with different adhesives | Baseline
  Restored teeth were evaluated according to FDI criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Karadaş, PhD, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Muhammet Karadaş, Rize, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No